CLINICAL TRIAL: NCT05694559
Title: Connecting Black Families in Houston, Texas to Hereditary Cancer Genetic Counseling, Genetic Testing, and Cascade Testing by Using a Simple Genetic Risk Screening Tool and Telegenetics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2022-0328; NCI-2023-00252 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms | interventions — Genetic Testing; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genetic Testing and Counseling (Experimental): Participants will be given a saliva collection kit to collect a saliva sample for hereditary cancer and genetic testing.
  Interventions: Behavioral: Genetic Testing and Counseling
- Screening Form (Experimental): Participants will complete a screening form to assess your risk of hereditary breast and colorectal cancers. You will be asked to provide your:
  * Name and contact information (including your address, phone number, and email)
  * Demographic information (including your age, race, and ethnicity)
  * Health insurance status
  * Annual household income
  * Personal and family history of cancer, including diagnosis and age at diagnosis
  Interventions: Behavioral: Screening Form

INTERVENTIONS:
Behavioral: Genetic Testing and Counseling — Participants will complete testing
  Arms: Genetic Testing and Counseling
Behavioral: Screening Form — Participants will complete forms with demographics and history
  Arms: Screening Form

SUMMARY:
To identify Black individuals who are eligible for genetic testing through trusted community organizations, and to connect Black individuals and their families to genetic testing and counseling so that they can know their cancer risk and how to decrease it.

DETAILED DESCRIPTION:
Primary Objectives:

* To identify 300 Black families, at least one individual per family, eligible for genetic testing using our validated simple genetic risk screening tool (GRST) 1, via collaboration with trusted community organizations. For individuals eligible for genetic testing, we will counsel them about genetic testing, including reviewing GRST results, explaining why they are eligible for genetic testing as part of standard-of-care, explaining what this entails, offering on-site or remote genetic testing, and explaining that they will be connected to a genetic counselor if they have a pathogenic mutation (PV) of a variant of unknown significance (VUS), including resources for family cascade genetic testing.
* To provide genetic testing to 150 Black individuals and families and provide genetic counseling and risk reduction resources to individuals with a PV or VUS, including cascade genetic testing for their family members.

ELIGIBILITY:
Inclusion Criteria:

* Any participant over 18 years old who self-identifies as Black or African-American and signs an informed consent form, also referred to as the 'Permission to Contact' form, to be part of our study.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
genetic risk screening tool (GRST) questionnaire | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Arun, MD, Principal Investigator — MD Anderson Cancer Cneter
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org